CLINICAL TRIAL: NCT05472116
Title: Capillary Refill Time Measurement Utilizing Mobile Application in Children
Acronym: CapApp
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: pending2
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Healthy Children (1 Month to 17 Years Old)
Keywords: Capillary Refill; Mobile Health Application; Pediatrics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Mobile Health application (CapApp) — Mobile Health application (CapApp) will be used to measure capillary refill time in a healthy pediatric population and compared to two additional manual methods to include both human and computer annotation and mobile health application (Cap App).

SUMMARY:
To determine the accuracy and precision of capillary refill time measurement using a mobile health application (Cap App) in a healthy pediatric population. This will be a cross-sectional study measuring the capillary refill time in a healthy pediatric population using both the Cap App and two additional manual methods which will serve as the comparison.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 1 month to 17 years

Exclusion Criteria:

* Fever or hypothermia
* Chronic illness including cardiovascular or renal disease
* Severe injury or blood loss
* Dehydration
* Raynaud's phenomenon

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children age 1 month to 17 years
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans on sharing results of the individual participant study data or aggregate study data with the participants. The data will be kept blinded from the research team members at the time of collection and, thus, no information will be shared with the participants.

RESULTS

PARTICIPANT FLOW:
Groups:
- Mobile Health Application: Mobile Health application (CapApp) will be used to measure capillary refill time in a healthy pediatric population and compared to two additional manual methods to include both human and computer annotation and mobile health application (Cap App).
Period: Overall Study
Arm/Group | Mobile Health Application
Started | 193
Completed | 152
Not Completed | 41

BASELINE CHARACTERISTICS:
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 152
  Between 18 and 65 years | 0
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 82
  Male | 69
  unreported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 114
  More than one race | 10
  Unknown or Not Reported | 16

OUTCOME MEASURES:

1. Primary Outcome: Accuracy and Precision of a Mobile Health Application (Cap App)
Description: Capillary refill time (CRT) of Cap App compared to two manual methods
Time Frame: Time it takes for blood to return to issue on the fingertip after pressure application for 5 seconds
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 152
seconds | 0.01 (1.31)

ADVERSE EVENTS:
Description: Data on adverse events was not collected
Arm/Group | Mobile Health Application
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT05472116/Prot_SAP_000.pdf